CLINICAL TRIAL: NCT01655420
Title: Patient-Reported Outcomes With LASIK: PROWL-2
Brief Title: Patient Reported Outcomes With LASIK: PROWL-2
Acronym: PROWL-2
Status: Completed | Type: Observational
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20112124
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Laser in Situ Keratomileusis
Keywords: Myopia; Hyperopia; Astigmatism; Patient-reported outcomes; Patient satisfaction; Refractive Error; Emmetropia; Dry eyes; Glare; Halos; Patient expectations
MeSH Terms: conditions — Myopia; Hyperopia; Astigmatism; Patient Satisfaction; Refractive Errors; Dry Eye Syndromes | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LASIK: Individuals aged 21 to 84 years planning to undergo refractive surgery using LASIK for myopia, hyperopia, or astigmatism
  Interventions: Procedure: LASIK

INTERVENTIONS:
Procedure: LASIK — Laser eye surgery
  Other Names: Refractive surgery using LASIK for myopia, hyperopia, or astigmatism

SUMMARY:
This study evaluates a questionaire designed to measure satisfaction and ophthalmic-related quality of life (QoL) of 300 civilian participants prior to and three months following state-of-the-art laser in situ keratomileusis (LASIK).

DETAILED DESCRIPTION:
The LASIK Quality of Life Collaboration Project (LQOLCP) is a government partnership among the FDA's Center for Devices and Radiological Health (CDRH), the Department of Defense, and the National Eye Institute (NEI). This project examines patient-reported outcomes (PROs) following LASIK surgery. This three-phased project is part of FDA's ongoing effort to better monitor and improve the safety and effectiveness of lasers used in LASIK surgery. PROWL-2 is the third phase of the larger LQOLCP project. The primary objective of PROWL-2 is to explore the psychometric properties of a computer-based questionnaire assessing the patient-reported outcomes of satisfaction and ophthalmic-related quality of life before and over a period of 3 months following LASIK. This questionnaire initially developed and examined in PROWL-1 (a military population) will be examined psychometrically in a civilian population. PROWL-2 is a prospective, multi-center, observational study in which a participant's pre-operative status will serve as the baseline for one-month and three-month post-surgical comparisons. Three hundred (300) participants planning to undergo refractive surgery using LASIK for myopia, hyperopia, or astigmatism will be enrolled in this study from five (5) clinical sites across the United States. Additionally, routine clinical data will be collected pre- and post-operatively (e.g., best corrected visual acuity, manifest refraction, wavefront aberrometry, conreal topography, and other clinical assessments) and questionnaires will be independently administered pre-operatively and at the one-month and three-month post-operative visits.

ELIGIBILITY:
Inclusion Criteria:

* Investigators will be instructed to base subject eligibility on the Professional Use Information for their specific laser and keratome system, including but not limited to subjects who:
* Are aged 21 years or older.
* Have the ability to give informed consent.
* Speak and read English fluently.
* Have not previously had any form of refractive surgery, including prior LASIK or cataract surgery.
* May benefit from increased spectacle independence.
* Have been determined to be a good candidate for the LASIK procedure based on the investigator's assessment of medical and ophthalmic health, general cognitive function, and physical and social limitations.
* Have a treatment target of bilateral emmetropia. Of note, an eye must be treated within 7 days of the fellow eye.
* Express willingness and potential ability to return for all follow-up examinations through the 3-month follow-up exam under the care of the treating investigator.
* Have access to a computer with internet service.

Ages: 21 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals age of 21 to 84 years planning to undergo refractive surgery using LASIK for myopia, hyperopia, or astigmatism
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-07

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Stanford University School of Medicine, Stanford, California
  - 20/20 Institute, Indianapolis, Indiana
  - Durrie Vision, Overland Park, Kansas
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Vance Thompson Vision, Sioux Falls, South Dakota

REFERENCES:
- [Result] Eydelman M, Hilmantel G, Tarver ME, Hofmeister EM, May J, Hammel K, Hays RD, Ferris F 3rd. Symptoms and Satisfaction of Patients in the Patient-Reported Outcomes With Laser In Situ Keratomileusis (PROWL) Studies. JAMA Ophthalmol. 2017 Jan 1;135(1):13-22. doi: 10.1001/jamaophthalmol.2016.4587. PMID 27893066
- [Result] Hays RD, Tarver ME, Spritzer KL, Reise S, Hilmantel G, Hofmeister EM, Hammel K, May J, Ferris F 3rd, Eydelman M. Assessment of the Psychometric Properties of a Questionnaire Assessing Patient-Reported Outcomes With Laser In Situ Keratomileusis (PROWL). JAMA Ophthalmol. 2017 Jan 1;135(1):3-12. doi: 10.1001/jamaophthalmol.2016.4597. PMID 27893063